CLINICAL TRIAL: NCT02434094
Title: Development of a Comprehensive AP Training Curriculum for Adults
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Sue Brown, Principal Investigator, University of Virginia
Other Study IDs: 18032
Record Dates: First submitted 2015-04-29; First posted 2015-05-05 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Assistant (DiAs); Continuous Glucose Monitor (CGM); Insulin Pump; Human Factors; Focus Group; Artificial Pancreas (AP); eDAPT (electronic Diabetes Artificial Pancreas Training)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- T1DM Clinicians: Clinicals currently teaching T1DM patients how to use insulin pumps and continuous glucose monitors will be asked to complete the eDAPT on-line training program.
  Interventions: Behavioral: eDAPT on-line training program
- T1DM Subjects with DiAs experience: T1DM subjects will prior DiAs experience will be asked to complete the eDAPT on-line training program.
  Interventions: Behavioral: eDAPT on-line training program
- T1DM Subjects with no prior DiAs experience: T1DM subjects will no prior DiAs experience will be asked to complete the eDAPT on-line training program.
  Interventions: Behavioral: eDAPT on-line training program

INTERVENTIONS:
Behavioral: eDAPT on-line training program — A series of modules used to train on the web based training system for the artificial pancreas (AP) prototype, DiAs.

SUMMARY:
An e-learning training program is to prepare people with diabetes and their physicians on the use of UVA's Artificial Pancreas prototype -- Diabetes Assistant (DiAs).

DETAILED DESCRIPTION:
This project will develop and test a comprehensive, web based training system for the artificial pancreas (AP) prototype identified as eDAPT (electronic Diabetes Artificial Pancreas Training). This e-learning training program is to prepare people with diabetes and their physicians on the use of UVA's Artificial Pancreas prototype -- Diabetes Assistant (DiAs), a software platform for the development and outpatient testing of smart phone based systems for Closed Loop Control of diabetes. The e-learning training program will be used in adjunct to in-person training with study staff at the onset of a clinical trial. It will be especially important as the number of clinical sites that use DiAs continue to grow both in the United States and internationally. It is also a critical step in moving the DiAs closer to a commercial product. A validated training program is required to proceed with the Food and Drug Administration (FDA) for both pivotal clinical trials and commercial approval of the AP.

ELIGIBILITY:
Diabetes Clinicians Inclusion Criteria:

* Endocrinologist, Certified Diabetes Educator, Nurse Practitioner actively managing patients with type 1 diabetes on insulin pumps and continuous glucose monitoring therapy
* Actively managing patients using insulin pumps for at least one year

Former & Novice Study Subjects Inclusion Criteria:

* Have Type 1 Diabetes Mellitus as defined by American Diabetes Association criteria or judgment of physician for at least 1 year
* No previous experience with the artificial pancreas system in a clinical trial
* Currently using insulin pump to manage their type 1 diabetes for at least one year
* Actively using an insulin pump with bolus calculator feature including predefined parameters for carbohydrate ratio, insulin sensitivity factor, target BG and active insulin
* Knowledge of continuous glucose monitors

Former Study Subjects Inclusion Criteria:

• Previous experience with the artificial pancreas system in a clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * clinicians who manage patients on insulin pumps and continuous glucose monitors
  * participants former study participants who have experience operating DiAs.
  * participants who wear an insulin pump and continuous glucose monitor but have no experience DiAs.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Validated eDAPT training tool | 2 hours
  Subjects learn how to properly operate & configure DiAs.
Human factors feedback | 2 hours
  Administration of knowledge tests and focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Sue Brown, MD, Principal Investigator — UVA Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States